CLINICAL TRIAL: NCT01272531
Title: Pharmacogenomics of Mood Stabilizer Response in Bipolar Disorder (PGBD)
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, John Kelsoe, Professor, University of California, San Diego
Other Study IDs: NIH 1 U01 MH92758-01; U01MH092758 (NIH)
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Bipolar Affective Disorder
Keywords: pharmacogenetics; bipolar disorders; affective disorders; mood disorders; pharmacologic actions; psychotropic drugs; antimanic agents; antidepressant agents; lithium; lithium carbonate; Lithobid; Eskalith; divalproex; divalproex sodium; Depakote; valproate
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders | interventions — Lithium Carbonate; Valproic Acid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from patients with bipolar disorder
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- lithium: All study subjects will be started on lithium and taken off other medications, such as antidepressants, antipsychotic or other mood stabilizers used to control their mood. They will be stabilized over a 3 month time period, observed for one month, the followed every 2 months for 2 years.
  Interventions: Drug: Mood stabilizer treatment
- valproate: Subjects that do not achieve stabilization or relapse while on lithium monotherapy will be started on valproate (VPA), in an identically designed prospective trial of VPA.
  Interventions: Drug: Mood stabilizer treatment

INTERVENTIONS:
Drug: Mood stabilizer treatment — lithium or valproate
  Other Names: lithium carbonate; Eskalith; Lithobid; divalproex sodium; Depakote; Depakene

SUMMARY:
This is a prospective pharmacogenomics study of mood stabilizer response. The goal of this work is to identify genes associated with good response of patients with bipolar disorder to two commonly used mood stabilizing agents, lithium and valproate.

DETAILED DESCRIPTION:
All subjects meeting study inclusion criteria will be started on lithium. Those that fail lithium will be crossed over to valproate (VPA). Those that also fail VPA will be again crossed-over to a standardized treatment as usual (TAU) arm. Subjects who are eligible for the study must be at least 18 years of age and have been diagnosed or are thought to have bipolar I disorder with at least one episode of mood instability in the last 12 months. They must also be eligible to take lithium and, if female and of child bearing age, agree to use adequate birth control methods and to inform their doctor of their plans to become pregnant.

ELIGIBILITY:
Inclusion Criteria:

* Any phase of bipolar I disorder including, depressive, manic, hypomanic, mixed, or baseline/euthymic/not symptomatic;
* Lithium naïve patients and inadequately past lithium treated patients will be required to have had at least one affective episode in the last 12 months meeting DSM-IV criteria. Current lithium treated patients (CLTPs) will be stable on lithium monotherapy and will be exempted from this criterion if they have had no mood episodes meeting DSM-IV criteria in the last 6 months;
* Both outpatients and inpatients will be permitted to enroll into this study;
* Able to give informed consent, in the judgment of the investigator;
* Age greater than or equal to 18 years;
* Women of child bearing potential agree to inform their doctor at the earliest possible time of their plans to conceive, and to use adequate contraception (e.g. oral contraceptives, intrauterine device, barrier methods, or total abstinence from intercourse), and to understand the risks of lithium to the fetus and infant. Depo Provera is acceptable if it is started 3 months prior to enrollment.

Exclusion Criteria:

* Unwilling or unable to comply with study requirements;
* Renal impairment (serum creatinine >1.5 mg/dL);
* Thyroid stimulating hormone (TSH) over >20% above the upper normal limit (participants maintained on thyroid medication must be euthyroid for at least 3 months before Visit 1;
* Other contraindication to lithium;
* Currently in crisis such that inpatient hospitalization or other crisis management should take priority;
* Subjects with alcohol/drug dependence who meet criteria for physical dependence requiring acute detoxification;
* Pregnant or breastfeeding;
* Women of child-bearing potential who aren't able to agree to the requirements specified above;
* Those who have participated in a clinical trial of an investigational drug within the past 1 month;
* Inability to agree to comply with the visit schedule or study procedures;
* History of lithium toxicity, not due to mismanagement or overdose that required treatment;
* Current unstable medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient and outpatients with bipolar affective disorder
Sampling Method: Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Time to relapse | every 2 months for 2 years
  Relapse definition:
  * meets criteria for mania and is considered "markedly ill" or worse; or
  * meets criteria for major depression with 4 week duration;
  * meets criteria for a mixed episode and is considered "markedly ill" or worse.

CONTACTS AND LOCATIONS:
Overall Officials: John R Kelsoe, M.D., Principal Investigator — University of California, San Diego
Locations (10):
- United States (8):
  - University of California San Diego, San Diego, California
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Dalhousie University, Halifax, Nova Scotia, Canada
- University of Bergen, Bergen, Norway

REFERENCES:
- [Derived] Oedegaard KJ, Alda M, Anand A, Andreassen OA, Balaraman Y, Berrettini WH, Bhattacharjee A, Brennand KJ, Burdick KE, Calabrese JR, Calkin CV, Claasen A, Coryell WH, Craig D, DeModena A, Frye M, Gage FH, Gao K, Garnham J, Gershon E, Jakobsen P, Leckband SG, McCarthy MJ, McInnis MG, Maihofer AX, Mertens J, Morken G, Nievergelt CM, Nurnberger J, Pham S, Schoeyen H, Shekhtman T, Shilling PD, Szelinger S, Tarwater B, Yao J, Zandi PP, Kelsoe JR. The Pharmacogenomics of Bipolar Disorder study (PGBD): identification of genes for lithium response in a prospective sample. BMC Psychiatry. 2016 May 5;16:129. doi: 10.1186/s12888-016-0732-x. PMID 27150464
- See also: PGBD website — http://www.lithium.ucsd.edu